CLINICAL TRIAL: NCT03589300
Title: Persona® TM Tibia Clinical Outcomes Study: Prospective Multicenter Study of the Persona® Trabecular Metal Tibia
Brief Title: Persona TM Tibia Clinical Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K.CR.I.G.16.33
Record Dates: First submitted 2018-06-20; First posted 2018-07-17 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis; Polyarthritis; Collagen Disorders and/or Avascular Necrosis of the Femoral Condyle; Post-traumatic Loss of Joint Configuration; Moderate Valgus, Varus, or Flexion Deformities
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Persona TM Tibia subjects (Other): Subjects that receive the Persona TM Tibia implant
  Interventions: Device: Persona TM Tibia

INTERVENTIONS:
Device: Persona TM Tibia — Trabecular Metal tibia used in primary cementless total knee arthroplasty

SUMMARY:
The primary objective of this study is to evaluate clinical performance for the commercially available Persona TM Tibia used in primary cementless tibia total knee arthroplasty.

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-randomized clinical study designed to facilitate the collection and evaluation of radiographic parameters, pain and function, survival of the device,and adverse event data.

The study will require each site to obtain IRB approval prior to study enrollment. All potential study subjects will be required to participate in the Informed Consent Process.

All study subjects will undergo preoperative clinical evaluations prior to their cementless tibia total knee arthroplasty. An immediate postoperative radiograph will be required. Postoperative clinical follow-up and radiographic evaluations will be conducted at 6 weeks, 6 months, 1 year, and 2 years.

The primary endpoint of this study is to evaluate the clinical performance of the implant at 2 years postoperatively using radiographic parameters. Radiographs will be assessed for the absence of progressive tibial radiolucencies, as defined in the radiographic protocol.

The secondary endpoints of this study will evaluate the clinical performance of the implant at 2 years postoperatively, based upon:

* No revisions for any reason
* Oxford Knee Score >38

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years of age.
2. Patient qualifies for a primary cementless tibia total knee arthroplasty based on physical exam and medical history, including diagnosis of severe knee pain and disability due to at least one of the following:

   1. Rheumatoid arthritis, osteoarthritis, traumatic arthritis, polyarthritis.
   2. Collagen disorders and/or avascular necrosis of the femoral condyle.
   3. Post-traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy.
   4. Moderate valgus, varus, or flexion deformities.
   5. The salvage of previously failed surgical attempts that did not include partial or total knee arthroplasty of the ipsilateral knee.
3. Patient has participated in the study-related Informed Consent process.
4. Patient is willing and able to provide written Informed Consent by signing and dating the IRB approved Informed Consent Form.
5. Patient is willing and able to complete scheduled study procedures and follow-up evaluations as described in the Informed Consent Form.
6. Independent of study participation, patient is a candidate for commercially available cementless Persona TM tibial knee component, implanted in accordance with product labeling.

Exclusion Criteria:

1. Previous history of infection in the affected joint.
2. Active local or systemic infection that may affect the prosthetic joint.
3. Insufficient bone stock on femoral or tibial surfaces.
4. Skeletal immaturity.
5. Neuropathic arthropathy.
6. Osteoporosis or any loss of musculature or neuromuscular disease that compromises the affected limb.
7. A stable, painless arthrodesis in a satisfactory functional position.
8. Severe instability secondary to the absence of collateral ligament integrity.
9. Rheumatoid arthritis accompanied by an ulcer of the skin or a history of recurrent breakdown of the skin.
10. Patient has previously received partial or total knee arthroplasty for the ipsilateral knee.
11. Patient is currently participating in any other surgical intervention studies or pain management studies.
12. Patient is known to be pregnant or considered a member of a protected population (e.g., prisoner, mentally incompetent, etc.).
13. Patient has a known or suspected sensitivity or allergy to one or more of the implant materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (7):
- United States (7):
  - LA BioMed at Harbor-UCLA Medical Center, Torrance, California
  - Cornerstone Orthopaedics & Sports Medicine, P.C., Wheat Ridge, Colorado
  - Hawaii Pacific Health, Honolulu, Hawaii
  - Henry County Orthopedics and Sports Medicine, New Castle, Indiana
  - Woods Mill Orthopedics, Ltd, Chesterfield, Missouri
  - Pinehurst Surgical Clinic, Pinehurst, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Knees
Groups:
- Persona TM Tibia: Persona Trabecular Metal (TM) Tibia used in primary cementless total knee arthroplasty
Period: Overall Study
Arm/Group | Persona TM Tibia
Started (125 participants (148 knees) proceeded with surgery and received the Persona TM Tibia implant (study device). There were 102 participants with surgery on one knee and 23 participants with surgery on both knees.) | 125; 148 Knees
Completed (102 participants (120 knees) completed the 2 year follow-up physical exam.) | 102; 120 Knees
Not Completed | 23; 28 Knees
Not completed — Adverse Event | 2
Not completed — Death | 4
Not completed — Lost to Follow-up | 12
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: Demographics are being reported for the 148 knees that received the Persona TM Tibia implant (study device).
Units Other Than Participants: Knees
Groups:
- Persona TM Tibia: Persona Trabecular Metal Tibia used in primary cementless total knee arthroplasty
Arm/Group | Persona TM Tibia
Number analyzed (Participants) | 125
Number analyzed (Knees) | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.28 (8.93)
Sex: Female, Male [Count of Units; unit: Knees]
  Female | 64
  Male | 84
Race/Ethnicity, Customized [Count of Units; unit: Knees]
  African American or Black | 9
  American Indian or Alaska Native | 1
  Asian | 16
  Hispanic or Latino | 21
  Native Hawaiian or Other Pacific Islander | 2
  White | 99
Region of Enrollment [Number; unit: Knees]
  United States | 148

OUTCOME MEASURES:

1. Primary Outcome: Radiograph Assessment of Progressive Tibial Radiolucencies
Description: Progressive tibial radiolucency will be derived in accordance with the following definitions:
  Absent: No evidence of an increase in either radiolucency extent (number of zones involved) or measured width within a zone.
  Present: Presence of either: An increase in the number of zones with a measured tibial radiolucency, OR an increase in the measured tibial radiolucency width within a zone of >0.5 mm.
  Unable to assess: One or more of the component factors necessary to derive progressive tibial radiolucency is unavailable.
Time Frame: 2 years
Population: 99 participants (117 knees) had radiographs analyzed at the 2 year follow-up interval.
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | Persona TM Tibia
Number analyzed (Participants) | 99
Number analyzed (Knees) | 117
Knees
  Absent | 110
  Present | 4
  Unable to assess | 3

2. Secondary Outcome: Oxford Knee Score
Description: The Oxford Knee Score is a patient completed 12 question metric to rate a patient's knee pain and function using an ordinal 0 - 4 point scale. The total score is obtained by calculating the sum of the 12 items. The maximum score is 48 points (best) and the minimum score is 0 points (worst).
Time Frame: 2 years
Population: 97 participants (115 knees) completed the Oxford Knee Score (OKS) at the 2 year follow-up interval.
  Literature suggests that Oxford Knee Scores above 41 are considered excellent and scores from 34 to 41 are considered good. The endpoint was designed to distinguish scores above 38.
  Reference: Murray et al. (2007). The use of the Oxford hip and knee scores. Bone & Joint Journal, 89(8), 1010-1014
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | Persona TM Tibia
Number analyzed (Participants) | 97
Number analyzed (Knees) | 115
Knees
  OKS >38 | 95
  OKS <=38 | 20

3. Secondary Outcome: Revision Rate
Description: Rate of the number of revisions for any reason
Time Frame: 2 years
Population: A revision is when the study implant is removed/revised due to an adverse event. Of the 148 knees that received the Persona TM Tibia implant, there were 2 reported revisions.
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | Persona TM Tibia
Number analyzed (Participants) | 125
Number analyzed (Knees) | 148
Knees
  Number of knees not revised | 146
  Number of knees revised | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant from the date of study device surgery through the 2 year follow-up interval. An exception is for the participants who did not complete the study, where adverse events were collected through the date of when the participant exited the study.
Arm/Group | Persona TM Tibia
All-Cause Mortality (participants affected / at risk) | 4/125
Serious Adverse Events (participants affected / at risk) | 15/125
Other Adverse Events (participants affected / at risk) | 69/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persona TM Tibia (N=125)
Cellulitis/Redness/Blistering (Skin and subcutaneous tissue disorders) | 1 (1) — Study knee related
Contralateral Knee Replacement (UKA or TKA) (Surgical and medical procedures) | 3 (3) — General adverse event (not study knee)
Deep Wound Infection (Infections and infestations) | 1 (1) — Study knee related
Effusion/Swelling/Edema (Musculoskeletal and connective tissue disorders) | 1 (1) — Study knee related
Endocrine (Endocrine disorders) | 1 (1) — General adverse event (not study knee)
Gastrointestinal (Gastrointestinal disorders) | 1 (1) — General adverse event (not study knee)
Hematological/Abnormal Lab (Blood and lymphatic system disorders) | 1 (1) — General adverse event (not study knee)
Infection (not study knee) (Infections and infestations) | 1 (1) — General adverse event (not study knee)
Musculoskeletal (not study knee) (Musculoskeletal and connective tissue disorders) | 5 (5) — General adverse event (not study knee)
Pain (progressive/persistent) (Musculoskeletal and connective tissue disorders) | 1 (1) — Study knee related
Traumatic Injury (not study knee) (Injury, poisoning and procedural complications) | 3 (3) — General adverse event (not study knee)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persona TM Tibia (N=125)
Cardiovascular (Cardiac disorders) | 6 (6) — General adverse event (not study knee)
Cellulitis/Redness/Blistering (Skin and subcutaneous tissue disorders) | 1 (1) — Study knee related
Clicking/Popping/Crepitus/Grinding (Musculoskeletal and connective tissue disorders) | 4 (4) — Study knee related
Contralateral Knee Replacement (UKA or TKA) (Surgical and medical procedures) | 6 (6) — General adverse event (not study knee)
Deep Wound Infection (Infections and infestations) | 1 (1) — Study knee related
Dermatological (Skin and subcutaneous tissue disorders) | 3 (3) — General adverse event (not study knee)
Effusion/Swelling/Edema (Musculoskeletal and connective tissue disorders) | 1 (1) — Study knee related
Endocrine (Endocrine disorders) | 3 (3) — General adverse event (not study knee)
Femoral Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 3 (3) — General adverse event (not study knee)
Genitourinary/Renal (Renal and urinary disorders) | 5 (5)
Hematological/Abnormal Lab (Blood and lymphatic system disorders) | 3 (3) — General adverse event (not study knee)
Infection (not study knee) (Infections and infestations) | 2 (2) — General adverse event (not study knee)
Musculoskeletal (not study knee) (Musculoskeletal and connective tissue disorders) | 31 (36) — General adverse event (not study knee)
Neurological (Nervous system disorders) | 4 (4) — General adverse event (not study knee)
Other General Adverse Event (General disorders) | 5 (5) — General adverse event (not study knee)
Other Ipsilateral Knee Related Adverse Event (Musculoskeletal and connective tissue disorders) | 3 (3) — Study knee related
Pain (progressive/persistent) (Musculoskeletal and connective tissue disorders) | 13 (13) — Study knee related
Patellar Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Study knee related
Psychological (Psychiatric disorders) | 2 (2) — General adverse event (not study knee)
Pulmonary/Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) — General adverse event (not study knee)
Stiffness/Limited ROM (progress/persistent) (Musculoskeletal and connective tissue disorders) | 10 (10) — Study knee related
Traumatic Injury (not study knee) (Injury, poisoning and procedural complications) | 3 (3) — General adverse event (not study knee)
Traumatic Injury (study knee) (Injury, poisoning and procedural complications) | 3 (3) — Study knee related
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 1 (1) — Study knee related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT03589300/Prot_SAP_000.pdf